CLINICAL TRIAL: NCT05919940
Title: Improved Muscle Metabolism by Combination of Muscle Activation and Protein Substitution: a Randomized, Outcome-assessor Blinded, Proof-of-concept Study (IMEMPRO)
Brief Title: Improved Muscle Metabolism by Combination of Muscle Activation and Protein Substitution ( IMEMPRO )
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Fresenius Kabi (Industry); University Medicine Greifswald (Other); Berlin Institute of Health (Other); Universitätsklinikum Ulm (Unknown); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stefan Schaller, MD, Full Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMEMPRO
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: ICU Acquired Weakness; Muscle Atrophy; Energy Malnutrition Protein; Quality of Life; Morphological and Microscopic Findings; Metabolic Disturbance
Keywords: Early Mobilization and high-protein nutrition
MeSH Terms: conditions — Muscular Atrophy; Protein-Energy Malnutrition; Morphological and Microscopic Findings | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): High protein substitution plus NMES and EM
  Interventions: Dietary Supplement: Dietary Supplement: additional substitution of protein; Device: Neuromuscular electrical stimulation; Other: Early Mobilization
- Control Group (No Intervention): Nutrition and mobilization are carried out according to standard of care.

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: additional substitution of protein — Day one (admission) no nutrition is applied.
  Protein target is increased as follows:
  * to a level of 1,2g/kg/d on day 1 after ICU admission
  * to a level of 1,4g/kg/d on day 2 after ICU admission
  * to a level of 1,6g/kg/d on day 3 after ICU admission
  * to a level of 1,8g/kg/d on day 4 after ICU admission
  * to a level of 2,0g/kg/d from day 5 onwoards
  Additional protein is given within 2 hours after mobilization respectively:
  * to 0,125g/kg/d on day 1 after ICU admission
  * to 0,2g/kg/d on day 2 after ICU admission
  * to 0,25g/kg/d on day 3 after ICU admission
  * to 0,3g/kg/d from day 4 after ICU admission onwoards
  Arms: Intervention
Device: Neuromuscular electrical stimulation — twice daily 60 minutes till day 28 or ICU discharge
  Arms: Intervention
Other: Early Mobilization — at least 20 minutes a day following the SOMS concept. Duration: till 28 day or ICU discharge
  Arms: Intervention

SUMMARY:
Intensive Care Unit Acquired Weakness (ICUAW) describes muscle weakness that occurs in around 40% of patients during an intensive care stay. The morbidity and mortality of these patients is significantly increased over a 5-year period. The aim of this study is to investigate the combined effect of early enteral high-protein nutrition and early muscle activation on muscle atrophy in critically ill patients.

The study will include 40 patients (20 intervention, 20 observation) with requirement for enteral nutrition at time of inclusion. In the intervention group the maximum possible level of mobilization is carried out and muscles are activated twice a day using neuromuscular electrical stimulation (NMES). The nutrition plan of the intervention group is based on the applicable guidelines for intensive care medicine with exception of increased protein intake. The control group receives therapy without deviating from the standard according of the DGEM guideline.

The study aims to show that the decrease in muscle mass is significantly less than in the control group (primary hypothesis) via ultrasound of the rectus femoris muscle and in case of given consent muscle biopsy. As secondary hypothesis it is examined whether the combination of early high protein intake and muscle activation improves muscle strength and endurance.

DETAILED DESCRIPTION:
Intensive Care Unit Acquired Weakness (ICUAW) describes the clinically diagnosed manifestation of a neuromuscular organ dysfunction. It develops in approximately 40% of all intensive care unit patients amounting to at least 1.2 million patients annually in Germany. All these patients face a broad range of sequeleae and an increased mortality up to 5 years after ICU discharge. A characteristic pathophysiological phenomenon is an early severe muscle atrophy reaching 10% during the first days after ICU admission.

The current preventative and therapeutic approach for ICUAW is a combination of targeted risk factor management as well as early activation of muscles, i.e. neuromuscular electrical stimulation (NMES) and early mobilization as they have been shown to counteract the muscle atrophy and mediate different outcome benefits such as shorter ICU stay.

Nutrition is a key element of our daily life. Protein intake has been shown to affect lean mass and muscle mass. Research into specific nutritional strategies to treat or prevent ICUAW are scarce and the combination with early muscle activation has not been adequately explored.

The study will include 40 patients (20 intervention, 20 observation) who were admitted to an intensive care unit within the last 48 hours. A basic requirement for inclusion is an indication for enteral (via the gastrointestinal tract) nutrition at time of inclusion. In the intervention group, the ability to mobilize is assessed daily and the maximum possible level of mobilization is carried out and additional muscles are activated twice a day using neuromuscular electrical stimulation (NMES). The nutrition plan of the intervention group is based on the applicable guidelines for intensive care medicine. In this study, protein intake is increased in the interventional group. The control group receives therapy without deviating from the standard according to the SOP and DGEM guideline: "Clinical nutrition in intensive care medicine" 2018.

The study aims to show that the decrease in muscle mass is significantly less than in the control group (primary hypothesis) via ultrasound of the rectus femoris muscle and muscle biopsy. As a second hypothesis it is examined whether the combination of early high protein intake and muscle activation improves muscle strength and endurance compared to the control group.

Further exploratory analyses will investigate changes in the skeletal muscle glycogen content, skeletal muscle histology, skeletal muscle gene expression, skeletal muscle protein level, as well as metabolomic changes in blood and urine.

An additional blood sample will be taken after 90 days as part of a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* critically ill adults (≥ 18 years of age)
* newly admitted to the ICU (<48h)
* mechanically ventilated, expected to remain for at least 72h
* enteral nutrition is feasible

Exclusion Criteria:

* a BMI > 30
* expected death or withdrawal of life-sustaining treatments
* prior neuromuscular disease (e.g. paresis, myopathies, neuropathies)
* injury or disease preventing neuromuscular electrical stimulation or early mobilization (e.g., elevated intracranial pressure, unstable spine)
* a pacemaker or other electronic implant
* allergy to components of NMES adhesive
* have been dependent during activities of daily living prior to the hospital admission
* a language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in cross sectional area (ΔCSA) of the rectus femoris | day 1 (study inclusion) and 14 days
  Change in muscle mass between study inclusion and study day 14; measured as change of the cross sectional area (ΔCSA) of the rectus femoris muscle via ultrasound.

SECONDARY OUTCOMES:
change in muscle thickness of the rectus femoris | day 1 (study inclusion) until 90-day Follow-up
  change in muscle thickness from study inclusion until 90-day follow-up, measured via ultrasound.
change in echogenicity of the rectus femoris | day 1 (study inclusion) until 90-day Follow-up
  change in echogenicity from study inclusion until 90-day follow-up, measured via ultrasound.
change of the pennation angle of the rectus femoris | day 1 (study inclusion) until 90-day Follow-up
  change of the pennation angle from study inclusion until 90-day follow-up, measured via ultrasound.
change of the muscle strength, measured by the Medical Research Council score (MRC-score) | day 1 (study inclusion) until 90-day Follow-up
  change of the muscle strength, measured by the Medical Research Council score (MRC-score) from study inclusion until 90-day follow-up
change of the muscle strength, measured by handgrip dynamometry | day 1 (study inclusion) until 90-day Follow-up
  change of the muscle strength, measured by handgrip dynamometry from study inclusion until 90-day follow-up
change in muscle endurance | up to 90 day follow up
  change in muscle endurance, measured by the 6-minute walking test up to 90-day follow-up
change in physical physical function | up to 90-day follow-up
  change in physical physical function, measured by the Short Physical Performance Battery up to 90-day follow-up
development of quality of life | up to 90-day follow-up
  development of quality of life, measured by the Short Form-36 up to 90-day follow-up
change in Skeletal muscle mass | day 1 (study inclusion) until 90-day Follow-up
  change in Skeletal muscle mass, measured with bioelectrical impedance analysis up to 90-day follow-up.
change in extracellular volume | day 1 (study inclusion) until 90-day Follow-up
  change in extracellular volume, measured by the Body impedance analysis
change in the REE (Resting Energy Expenditure) | day 1 (study inclusion) until 90-day Follow-up
  change in the REE (Resting Energy Expenditure), measured by indirect calorimetry
urea-to-creatinine ratio | day 1 (study inclusion) until 90-day Follow-up
  urea-to-creatinine ratio from blood sample
Identify possible predictors of muscle wasting in urine metabolomics at ICU admission | day 1 (study inclusion) until 90-day Follow-up
  Among the urine metabolomics that will be measured, identify metabolites or combinations of metabolites whose high or low concentration(s) at ICU admission associate(s) with the amount of muscle loss. These metabolites are candidate biomarkers that could be used to identify individuals at risk of large muscle wasting and may give further insights into the mechanisms of muscle wasting.
Identify possible predictors of muscle wasting in the blood metabolome at ICU admission | day 1 (study inclusion) until 90-day Follow-up
  Among the blood metabolome that will be measured, identify metabolites or combinations of metabolites whose high or low concentration(s) at ICU admission associate(s) with the amount of muscle loss. These metabolites are candidate biomarkers that could be used to identify individuals at risk of large muscle wasting and may give further insights into the mechanisms of muscle wasting.

OTHER OUTCOMES:
in-hospital mortality | until 90-day Follow-up
  Mortality during the Hospital stay
Hospital LOS | until 90-day Follow-up
  Length of stay in the hospital
ICU-LOS | until 90-day Follow-up
  Length of stay in the ICU
Hospital mortality | until 90-day Follow-up
  Mortality during Hospital stay
Duration of Mechanical ventilation | until 90-day Follow-up
  Duration of invasive mechanical ventilator dependency
ICU mortality | until 90-day Follow-up
  Mortality during ICU stay
enzyme function in the rectus femoris | according to biopsy inbetween day 1-7
  Spectrophotometry will be done in muscle samples. All samples will be screened for influence of Intensive Care Unit Acquired Weakness (ICUAW) and correlation with blood metabolome changes.
protein content in the rectus femoris | according to biopsy inbetween day 1-7
  Western Blot will be done in muscle samples. All samples will be screened for influence of Intensive Care Unit Acquired Weakness (ICUAW) and correlation with blood metabolome changes.
geneexpression in the rectus femoris | according to biopsy inbetween day 1-7
  qPCR (quantitive polymerase chain reaction) will be done in muscle samples. All samples will be screened for influence of Intensive Care Unit Acquired Weakness (ICUAW) and correlation with blood metabolome changes.
Muscle morphology of the rectus femoris | according to biopsy inbetween day 1-7
  Light-and Electron-Microscopy will be done in muscle samples. All samples will be screened for influence of Intensive Care Unit Acquired Weakness (ICUAW) and correlation with blood metabolome changes.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Medical University of Vienna & Charité - Universitätsmedizin Berlin
Locations (4):
- Medical University of Vienna, Vienna, Vienna, Austria
- Germany (3):
  - Klinikum rechts der Isar, School of Medicine, Technical Universtity of Munich, Munich, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data can be requested on reasonable scientific request and data sharing contract, if necessary.
Supporting Information: Study Protocol, ICF
Time Frame: After publication of scientific manuscript.
Access Criteria: Deidentified data can be requested on reasonable scientific request and data sharing contract, if necessary.